CLINICAL TRIAL: NCT05302232
Title: Randomised Trial of Intra-articular Injection of Lidocaine Versus Placebo in Inflammatory Arthritis
Brief Title: Intra-articular Injection of Lidocaine in Inflammatory Arthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 311106
Record Dates: First submitted 2022-01-11; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-01

CONDITIONS: Inflammatory Arthritis
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Intervention Model Description: Patients will be randomised to receive joint injection of either lidocaine plus steroid or, as a control, just steroid injection
Who Masked: Participant
Masking Description: Treatment allocation will be single blinded, in that the researcher will know what intervention the patient is receiving but the patient will not.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine plus steroid (Experimental)
  Interventions: Diagnostic Test: depomedrone 40mg/ml + 1% lidocaine; Other: painDETECT questionnaire
- Steroid only (Placebo Comparator)
  Interventions: Diagnostic Test: depomedrone 40mg/ml+ 0.9% saline; Other: painDETECT questionnaire

INTERVENTIONS:
Diagnostic Test: depomedrone 40mg/ml + 1% lidocaine — Response to intra-articular injection of lidocaine as a diagnostic marker of peripheral pain
  Arms: Lidocaine plus steroid
Diagnostic Test: depomedrone 40mg/ml+ 0.9% saline — Response to intra-articular injection of steroid only as a placebo
  Arms: Steroid only
Other: painDETECT questionnaire — painDETECT questionnaire

SUMMARY:
To assess the contributions of peripheral neurons to joint pain, the investigators plan to ask patients to rate the pain in their chosen joint before and after an injection of local anaesthetic (lidocaine) and steroid into their joint. Lidocaine blocks voltage gated sodium channels (VGSCs) leading to a reversible block of action potential propagation in peripheral nerves. If the pain intensity reduces significantly following lidocaine injection, it suggests that the patients' pain is due to peripheral sensitization, and that this is dampened by the local anaesthetic. If the pain intensity does not change or only falls slightly, then other centrally mediated factors are contributing to pain.

Before the investigators can use this method, the investigators need to ensure that reductions in pain score following joint injection are not due to placebo effect. Therefore, as part of this validation study patients will be randomised to receive either lidocaine plus steroid or, as a control, just steroid injection. The steroid is the main part of therapy as it relieves inflammation over a prolonged period, but is slower acting than lidocaine, and should not have an effect within ten minutes. Any improvement in ranking of pain within 10 minutes by patients receiving just steroid will therefore be due to placebo effect. The investigators hypothesis is that there will be a significant difference in change in pain score before and after injection between the study group (lidocaine plus steroid) and control group (0.9% saline plus steroid). This will confirm the absence of a significant placebo effect and mean the differences in change in pain scores seen in the study group are due to differences in pain processing

DETAILED DESCRIPTION:
Patients will be randomised to receive joint injection of either lidocaine plus steroid or, as a control, just steroid injection. Pain scores (visual analogue score 0-10) in the chosen joint will be collected prior to injection and at 3, 5 and 10 minutes post injection. Pain scores will then again be collected at 1 month and 3 months to determine whether lidocaine reduced peripheral pain long term.

Intra-articular joint injection with steroids is a frequent procedure in usual care and the investigators will only perform this test when a joint injection +/- aspiration is clinically indicated. Use of lidocaine in addition to steroid injection varies between rheumatologists, with 50% of Guys' and St Thomas' Hospital rheumatologists routinely using lidocaine and steroid, and others giving steroid alone. Therefore, all patients will still receive the same intervention they would if they were not taking part in the study, the only difference is measurement of pain scores before and after.

In addition to collection of pain scores, the investigators will collect patient demographics and painDETECT questionnaire, a screening questionnaire which has been validated to identify neuropathic elements of pain in patients with IA.

The investigators hypothesis is that there will be a significant difference in change in pain score before and after injection between the study group (lidocaine plus steroid) and control group (0.9% saline plus steroid). This will confirm the absence of a significant placebo effect and mean the differences in change in pain scores seen in the study group are due to differences in pain processing.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of peripheral inflammatory joint disease
* Reporting current NRS pain ≥3 on a 0-10 scale
* Only perform this test when an aspiration and joint injection is clinically indicated and would be given as part of routine care

Exclusion Criteria:

* Under 18 years of age
* Unable or unwilling to provide informed written consent
* Unable to comply with study protocols
* Pregnancy and breastfeeding
* If the chosen joint has been aspirated or injected in the preceding 3 months
* Presence of joint damage in chosen joint as assessed by Professor Kirkham on x-ray of the chosen joint (as joint damage itself can stimulate peripheral nociceptors)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-04-18 (Estimated); Primary Completion 2022-10-18 (Estimated); Study Completion 2022-10-18 (Estimated)

PRIMARY OUTCOMES:
pain score 5 minutes post-injection | 5 minutes
  Visual analogue pain score 0-10

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Kirkham, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rutter-Locher Z, Norton S, Denk F, McMahon S, Taams LS, Kirkham BW, Bannister K. A randomised controlled trial of the effect of intra-articular lidocaine on pain scores in inflammatory arthritis. Pain. 2024 Nov 1;165(11):2578-2585. doi: 10.1097/j.pain.0000000000003291. Epub 2024 Jun 17. PMID 38888846